CLINICAL TRIAL: NCT01482390
Title: A Phase II, Randomized, Double-Blind, Multicenter, Parallel Group Study to Evaluate the Sustained Virologic Response of the HCV Polymerase Inhibitor Prodrug RO5024048 in Combination With Telaprevir and Pegasys®/Copegus® in Patients With Chronic Hepatitis C Genotype 1 Virus Infection Who Were Prior Null Responders to Treatment With Pegylated Interferon/Ribavirin
Brief Title: A Study of Mericitabine in Combination With Telaprevir and Peginterferon Alfa-2a / Ribavirin in Participants With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NV27779; 2011-002715-28 (EudraCT Number)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; 2'-fluoro-2'-methyl-3',5'-diisobutyryldeoxycytidine; peginterferon alfa-2a; telaprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- TVR (12 Weeks), MCB (24 Weeks), PEG-IFN/RBV (24 Weeks) (Experimental): Twelve weeks of therapy with MCB, TVR, and PEG-IFN/RBV, followed by 12 weeks of therapy with MCB and PEG-IFN/RBV (total treatment duration of 24 weeks).
  Interventions: Drug: Ribavirin; Drug: Mericitabine; Drug: Peginterferon Alfa-2a; Drug: Telaprevir
- TVR (12 Weeks), MCB (24 Weeks), PEG-IFN/RBV (48 Weeks) (Experimental): Twelve weeks of therapy with MCB, TVR, and PEG-IFN/RBV, followed by 12 weeks of therapy with MCB and PEG-IFN/RBV and then 12 weeks of therapy with PEG-IFN/RBV (total treatment duration of 48 weeks).
  Interventions: Drug: Ribavirin; Drug: Mericitabine; Drug: Peginterferon Alfa-2a; Drug: Telaprevir
- TVR, MCB, Placebo MCB( each for 12Weeks),PEG-IFN/RBV(48 Weeks) (Experimental): Twelve weeks of therapy with MCB, TVR, and PEG-IFN/RBV, followed by 12 weeks of therapy with placebo matching to MCB and PEG-IFN/RBV, and then 24 weeks of therapy with PEG-IFN/RBV (total treatment duration of 48 weeks).
  Interventions: Drug: Ribavirin; Drug: Mericitabine; Drug: Peginterferon Alfa-2a; Drug: Placebo; Drug: Telaprevir
- TVR(12 Weeks), Placebo MCB (24 Weeks), PEG-IFN/RBV(48 Weeks) (Active Comparator): Twelve weeks of therapy with placebo matching to MCB, TVR, PEG-IFN/RBV, will be followed by 12 weeks of therapy with placebo matching to MCB along with PEG-IFN/RBV , following 24 weeks of therapy with PEG-IFN/RBV (total treatment duration of 48 weeks).
  Interventions: Drug: Ribavirin; Drug: Peginterferon Alfa-2a; Drug: Placebo; Drug: Telaprevir

INTERVENTIONS:
Drug: Ribavirin — Participants will receive a total daily dose of 1000 milligrams (mg) (for participants weighing less than [<] 75 kg) or 1200 mg (for participants weighing greater than or equal to [>=] 75 kg) orally for 24 or 48 weeks.
  Other Names: Copegus
Drug: Mericitabine — Participants will receive mericitabine 1000 mg orally twice daily.
  Arms: TVR (12 Weeks), MCB (24 Weeks), PEG-IFN/RBV (24 Weeks); TVR (12 Weeks), MCB (24 Weeks), PEG-IFN/RBV (48 Weeks); TVR, MCB, Placebo MCB( each for 12Weeks),PEG-IFN/RBV(48 Weeks)
Drug: Peginterferon Alfa-2a — Participants will receive 180 micrograms (mcg) subcutaneous injection once weekly.
  Other Names: Pegasys
Drug: Placebo — Participants will receive placebo matching to mericitabine orally twice daily.
  Arms: TVR(12 Weeks), Placebo MCB (24 Weeks), PEG-IFN/RBV(48 Weeks); TVR, MCB, Placebo MCB( each for 12Weeks),PEG-IFN/RBV(48 Weeks)
Drug: Telaprevir — Participants will receive telaprevir 750 mg orally three times daily.

SUMMARY:
This randomized, double-blind, multi-center, parallel-group study will evaluate the sustained virologic response and the safety of mericitabine (RO5024048) (MCB) in combination with telaprevir (TVR) and peginterferon Alfa-2a (PEG-IFN) / ribavirin (RBV) in participants with chronic Hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C infection for at least 6 months duration
* Hepatitis C genotype 1a or 1b
* Participants must have discontinued prior hepatitis C treatment at least 12 weeks prior to enrollment in this study
* Participants showed a previous null response to therapy as defined by < 2 logarithm to the base 10 (log10) international units per milliliter (IU/mL) decrease in viral titer after at least 12 weeks of treatment with PEG-IFN/RBV

Exclusion Criteria:

* Hepatitis C infection with a genotype other than genotype 1a or 1b
* Body mass index < 18 or >= 36 kilograms per square meters (kg/m^2)
* Hepatitis A, hepatitis B, or human immunodeficiency virus (HIV) infection
* Herbal remedies <=1 month prior to the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
Percent of Participants With Sustained Virological Response 12 Weeks After End of Treatment (SVR12), as Determined by Polymerase Chain Reaction (PCR) Using Roche COBAS TaqMan Hepatitis C Virus (HCV) Test | 12 weeks after end of treatment (up to Week 60)

SECONDARY OUTCOMES:
Percentage of Participants With Sustained Virological Response 4 Weeks After End of Treatment (SVR-4), as Determined by PCR Using Roche COBAS TaqMan HCV Test | 4 weeks after end of treatment (up to Week 52)
Percentage of Participants With Sustained Virological Response 24 Weeks After End of Treatment (SVR-24), as Determined by PCR Using Roche COBAS TaqMan HCV Test | 24 weeks after end of treatment (up to Week 72)
Percentage of Participants With Virological Response Over Time From Week 2 to Week 48, as Determined by PCR Using Roche COBAS TaqMan HCV Test | Weeks 2, 4, 12, 24, and 48
Percentage of Participants With Treatment- Resistant Mutations, as Determined Using Standard Sequencing Technology | Baseline up to Week 60
Change From Baseline in HCV Ribonucleic Acid (RNA) Levels | Baseline, Weeks 1, 2, 4, 8, 12, 16, 20, 24, 30, 36, 42, 48, 52, 60, and 72
Percentage of Participants With Adverse Event | Baseline up to Week 72
Trough Concentration of RO4995855 (Parent Drug of Mericitabine) | Pre-dose (-0.5 hour) on Day 1 and Week 8; 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hour post dose in Week 8
Trough Concentration of Metabolite of RO4995855 (RO5012433) | Pre-dose (-0.5 hour) on Day 1 and Week 8; 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hour post dose in Week 8
Trough Concentration of Telaprevir | Pre-dose (-0.5 hour) on Day 1 and Week 8; 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12 hour post dose in Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- United States (15):
  - Birmingham Gastro Associates, P.C., Birmingham, Alabama
  - VA Long Beach Healthcare System, Long Beach, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - UCSD Antiviral Research Center, San Diego, California
  - Yale University, New Haven, Connecticut
  - Gastroenterology Group of Naples, Naples, Florida
  - John Hopkins Hospital, Lutherville, Maryland
  - Metrowest Medical Center, Framingham, Massachusetts
  - Saint Louis University Gastroenterology & Hepatology; Clinical Research Unit, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Carolina'S Center For Liver Disease, Statesville, North Carolina
  - Uni of Cincinnati College of Medicine; Div. of Digestive Diseases, Cincinnati, Ohio
  - Baylor Uni Medical Center; Division Of Hepatology/Transplantation; Annette C. and Harold C. Simmons, Dallas, Texas
  - McGuire; Veteran Affairs Med Ctr, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
- Canada (7):
  - Gordon & Leslie Diamond Health Care Centre; Dept. of Medicine - Division of Gastroenterology, Vancouver, British Columbia
  - GI Research Institute; Gastroenterology & Hepatology, Vancouver, British Columbia
  - Percuro Clinical Research Ltd., Victoria, British Columbia
  - Winnipeg Regional Health Authority; Section of Hepatology, Winnipeg, Manitoba
  - University Health Network - Toronto Western Hospital; Hepatology, Toronto, Ontario
  - Toronto Digest. Disease Asso., Woodbridge, Ontario
  - McGill University, Montreal Chest Institute; Viral and other Infectious, Montreal, Quebec
- France (3):
  - Hopital Claude Huriez;Gastro Enterologie, Lille
  - Fondation Hopital Saint Joseph; Gastro-Enterologie, Marseille
  - Hopital Purpan;Gastro Enterologie Hepatologie, Toulouse
- Germany (3):
  - Klinik Johann Wolfgang von Goethe Uni; Zentrum der Inneren Medizin; Medizinische Klinik I, Frankfurt am Main
  - Uniklinik Freiburg; Abteilung Innere Medizin II, Freiburg im Breisgau
  - Universitäts Klinikum; Schleswig-Holstein Kiel, Kiel
- Italy (3):
  - UNI DEGLI STUDI - POLICLINICA S. ORSOLA; Dipartimento Malattie dell'Apparato Digerente e Medicina In, Bologna, Emilia-Romagna
  - ASST GRANDE OSPEDALE METROPOLITANO NIGUARDA; Divisione Malattie Infettive, Milan, Lombardy
  - Ospedale Cisanello - Az. Osp. Pisana; Unità Operativa Di Gastroenterologia Ed Epatologia, Pisa, Tuscany
- Spain (4):
  - Hospital Universitario de Canarias; Servicio de Digestivo, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitari Vall d'Hebron; Departamento de Enfermedades Infecciosas, Barcelona
  - Hospital Clinic I Provincial; Servicio de Digestivo, Barcelona
  - Hospital Carlos III; Laboratorio de Biologia Molecular, Madrid
- United Kingdom (4):
  - Royal Bournemouth Hospital, Gastroenterology, Dorset
  - King'S College Hospital; Institute of Liver Studies, London
  - St George's Hospital, London
  - Imperial College Healthcare NHS Trust; Hepatology Clinical Research Facility, London

REFERENCES:
- [Derived] Wedemeyer H, Forns X, Hezode C, Lee SS, Scalori A, Voulgari A, Le Pogam S, Najera I, Thommes JA. Mericitabine and Either Boceprevir or Telaprevir in Combination with Peginterferon Alfa-2a plus Ribavirin for Patients with Chronic Hepatitis C Genotype 1 Infection and Prior Null Response: The Randomized DYNAMO 1 and DYNAMO 2 Studies. PLoS One. 2016 Jan 11;11(1):e0145409. doi: 10.1371/journal.pone.0145409. eCollection 2016. PMID 26752189